CLINICAL TRIAL: NCT00061243
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of a Multi-Gene, Polyvalent HIV-1 DNA Plasmid Prime/Env Protein Boost Vaccine Formulation, DP6-001 in Healthy Volunteers
Brief Title: Safety of and Immune Response to Polyvalent HIV-1 Vaccine in HIV Uninfected Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Jeff Kennedy, MD, University of Massachusetts School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N01AI05394; N01-AI05394
Record Dates: First submitted 2003-05-22; First posted 2003-05-23 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2005-12

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; DNA prime; Protein boost; HIV Seronegativity; HIV preventive vaccine
MeSH Terms: conditions — HIV Infections

ARMS (5):
- 1 (Experimental): Participants will receive different doses of the vaccine to determine the optimal dose
  Interventions: Biological: HIV-1 DNA vaccine with protein vaccine boost
- 2 (Experimental): Participants will receive different doses of the vaccine to determine the optimal dose
  Interventions: Biological: HIV-1 DNA vaccine with protein vaccine boost
- 3 (Experimental): Participants will receive different doses of the vaccine to determine the optimal dose
  Interventions: Biological: HIV-1 DNA vaccine with protein vaccine boost
- 4 (Experimental): Participants will receive the vaccine through either intradermal or intramuscular administration
  Interventions: Biological: HIV-1 DNA vaccine with protein vaccine boost
- 5 (Experimental): Participants will receive the vaccine through either intradermal or intramuscular administration
  Interventions: Biological: HIV-1 DNA vaccine with protein vaccine boost

INTERVENTIONS:
Biological: HIV-1 DNA vaccine with protein vaccine boost — Three doses of DNA vaccination will be administered at weeks 0, 4, and 12, and 2 doses of protein vaccination at weeks 20 and 28

SUMMARY:
This study will evaluate the safety of and immune response to a new HIV vaccine. The vaccine in this trial uses pieces of HIV DNA and HIV proteins. The vaccine itself cannot cause HIV infection or AIDS.

DETAILED DESCRIPTION:
Unlike other viruses for which effective vaccines have been developed, HIV-1 has evolved mechanisms to evade immune control over virus replication. These mechanisms include the extraordinary genetic diversity of the virus, viral latency, and targeting of the immune system. Evolutional variations of the envelope gene have not only resulted in the development of different groups (M, N, and O) and subgroups (clades) in diverse geographic regions of the world, but also significant genomic variations within clades. These clade variants of HIV will require novel vaccine approaches to elicit population-based protective immunity. Viral latency is the ability of the virus to remain dormant for long periods through integrating its viral DNA into the host genome. Viral latency requires vaccines to produce immune response that are robust enough to kill the virus and that can be maintained over extended periods of time to produce lasting immunity. Finally, HIV-1 targets CD4 cells and thus compromises the immune surveillance mechanisms critical to maintaining both cellular and humoral immunity to HIV-1. Therefore, an effective vaccine against HIV-1 must bolster the development of broadly reactive neutralizing antibodies against genetic variants of HIV-1, as well as induce an effective HIV-specific CTL response to eliminate virus-infected cells. The ideal vaccine approach will produce long-term responses within these arms of host immunity. This study is designed to evaluate the safety, tolerability, and immunogenicity of a novel prophylactic vaccine consisting of DNA priming followed by a protein boost.

The first vaccine component administered in this study is a DNA vaccination; the second component is a recombinant protein vaccination. This combination will be used to determine whether the vaccine strategy can induce a balanced humoral and cell mediated immune responses to HIV-1.

Two HIV antigens, Gag and Env, are included in this study's vaccine formulation. Studies have shown that HIV-1 Gag is a potent inducer of cell mediated immune responses, while Env is the target of neutralizing antibody responses. The vaccine used in this study contains a 5-valent Env design (Env derived from one of 5 clades of HIV) in order to examine if a polyvalent Env formulation may expand the breadth of neutralizing antibody responses induced in human volunteers. For both DNA priming and protein boosting, a set of Env antigens from clades A, B, C, and E of HIV-1 M group will be produced (2 Env antigens from clade B and 1 Env each from the other three clades). All 5 Env antigens are selected from the primary HIV-1 viral isolates with the hope of producing broad antibody responses against the primary viruses circulating in the worldwide human population.

Thirty-six healthy volunteers will be randomized to one of five groups. Groups 1, 2, and 3 will receive different doses of the vaccine to determine the optimal dose. Groups 4 and 5 will receive the vaccine through either intradermal or intramuscular administration. Each group will receive 3 doses of DNA vaccination at weeks 0, 4, and 12, and 2 doses of protein vaccination at weeks 20 and 28. Blood sampling throughout the duration of the study will provide an assessment of the safety and immunogenicity of the vaccine in healthy volunteers. It is expected that volunteers will be enrolled in this study for 1 year.

ELIGIBILITY:
Inclusion Criteria

* HIV uninfected
* Good general health as determined by medical history, physical examination, vital signs, and clinical laboratory measurements
* Body Mass Index (BMI) =< 32
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive
* Low risk for HIV exposure
* No co-existent endocrine conditions
* No evidence of hepatic insufficiency, significant renal insufficiency, or proteinuria
* Acceptable methods of contraception
* Anticipated availability for the planned follow-up period of one year

Exclusion Criteria

* Certain medications during the 2 weeks prior to study entry
* Donation of a unit of blood within 2 months prior to study entry
* Participation in a study of investigational or marketed drugs within 1 month prior to study entry
* Blood transfusion within 6 months prior to study entry
* Pregnant, breastfeeding, or planning pregnancy during the study period
* History of significant adverse reaction to any vaccine
* Prior receipt of any experimental HIV vaccine
* Morbid obesity (> 195% of ideal body weight)
* Hypertension (patients may be taking concomitant antihypertensive medication during the study if approved by study officials)
* History of chronic medical illness, malignancy, or autoimmune disorder
* History of immunodeficiency or treatment with immunosuppressive medications
* History of organ transplant
* Medical or psychiatric obstacle to compliance with protocol
* Significant urine concentration of any drug that could interfere with the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2005-04 (Actual); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Throughout study

SECONDARY OUTCOMES:
Cross-clade neutralizing antibody | Throughout study
Cellular immunity | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Kennedy, MD, Study Director — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts School of Medicine, Worcester, Massachusetts, United States